CLINICAL TRIAL: NCT00310947
Title: Impact of Patient-Prosthesis-Mismatch and Aortic Valve Design on Coronary Flow Reserve Following Aortic Valve Replacement
Brief Title: Impact of Patient-Prosthesis-Mismatch on Coronary Flow Reserve
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Medtronic (Industry)
Other Study IDs: Coronary flow reserve
Record Dates: First submitted 2006-03-31; First posted 2006-04-05 (Estimated); Last update posted 2006-04-05 (Estimated); Status verified 2003-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Coronary flow reserve; Heart failure; prospective randomised
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
Complete normalization of CFR following AVR for aortic stenosis was observed only for stentless valves. Besides the superior hemodynamic performance this might explain the excellent long term results of this valve design.

ELIGIBILITY:
Inclusion Criteria:

Aortic valve stenosis

Exclusion Criteria:

Coronary artery disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2005-03; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kleine, MD,PhD, Principal Investigator — JW Goethe University Ffm
Locations (1):
- JW Goethe University Ffm, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Derived] Bakhtiary F, Schiemann M, Dzemali O, Dogan S, Schachinger V, Ackermann H, Moritz A, Kleine P. Impact of patient-prosthesis mismatch and aortic valve design on coronary flow reserve after aortic valve replacement. J Am Coll Cardiol. 2007 Feb 20;49(7):790-6. doi: 10.1016/j.jacc.2006.10.052. Epub 2007 Feb 5. PMID 17306709